CLINICAL TRIAL: NCT00729833
Title: Phase 1, Open Label, Sequential Cohort, Dose Escalation Study Of CP-751,871 In Combination With Sunitinib In Patients With Advanced Solid Tumors
Brief Title: Study Of CP-751,871 In Combination With Sunitinib In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021024
Record Dates: First submitted 2008-07-30; First posted 2008-08-08 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Cancer; Advanced Solid Tumors
MeSH Terms: interventions — figitumumab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-751,871 + Sunitinib (Experimental): Escalating cohorts of CP-751,871 + Sunitinib
  Interventions: Drug: CP-751,871; Drug: Sunitinib

INTERVENTIONS:
Drug: CP-751,871 — CP-751,871 IV, every 3 weeks
Drug: Sunitinib — Sunitinib - daily dosing

SUMMARY:
The study is being conducted to determine the maximum tolerated dose, overall safety and tolerability profile, and pharmacokinetic profile of CP-751,871 and sunitinib when given in combination with advanced solid tumors.

DETAILED DESCRIPTION:
The study was closed to enrollment on 14 Jan 2011 and terminated secondary to excessive screen failure rate and for business reasons associated with Pfizer's business decision to stop development of the figitumumab compound. Safety concerns did not contribute to the decision to terminate this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumors relapsed or refractory to standard therapy or for whom no standard therapy exists.
* ECOG Performance Status of 0 or 1;
* Total IGF-1 level ≥100 ng/ml;
* ECOG Performance Status of 0 or 1
* Adequate bone marrow, renal, and hepatic function

Exclusion Criteria:

* Concurrent treatment with any antitumor agents with the exception of LHRH agnosits for prostate cancer patients
* Treatment with any other investigational therapy within 4 weeks prior to study treatment
* Major surgery within 4 weeks of study treatment
* Prior treatment that may increase the risk of cardiac complications
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade 2 or greater
* Significant active cardiac disease, including hypertension that cannot be controlled by medications
* Greater than three (3) prior lines of cytotoxic therapy;
* Active infection
* Prior IGF-IR targeted therapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021024&StudyName=%20Study%20Of%20CP-751%2C871%20In%20Combination%20With%20Sunitinib%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab 10 mg/kg + Sunitinib 25 mg CDD: Figitumumab (CP-751,871) 10 milligram/kilogram (mg/kg) intravenous (IV) on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle on a continuous daily dosing (CDD) schedule. Dose escalation proceeded to the next cohort if 0/3 or 1/6 participant experienced a dose-limiting toxicity (DLT).
- Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD: Figitumumab 10 mg/kg IV on Day 1 of each 3-week cycle plus sunitinib 37.5 mg oral capsule on Day 1 of each 3-week cycle on a continuous daily dosing (CDD) schedule, until disease progression or unacceptable toxicity.
- Figitumumab 20 mg/kg + Sunitinib 25 mg CDD: Figitumumab 20 mg/kg IV on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle on a continuous daily dosing (CDD) schedule, until disease progression or unacceptable toxicity.
- Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1: Figitumumab 20 mg/kg on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle with 2 weeks of continuous daily dosing followed by 1 week off, until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Started | 20 | 7 | 12 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 20 | 7 | 12 | 6
Not completed — Death | 5 | 1 | 3 | 5
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 3 | 0
Not completed — Unspecified Reasons | 11 | 5 | 5 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All enrolled participants who received at least 1 dose of figitumumab plus sunitinib.
Groups:
- Figitumumab + Sunitinib (All Combined): All participants who received at least one dose of figitumumab plus sunitinib.
Arm/Group | Figitumumab + Sunitinib (All Combined)
Number analyzed (Participants) | 45
Age, Customized [Number; unit: participants]
  18 to 44 years | 11
  45 to 64 years | 22
  Greater than or equal to (>=) 65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: Number of participants with treatment-related Grade 3/4 toxicities that occurred during the defined time frame or that resulted in greater than or equal to (>=) 7 days delay in administration of Cycle 2.
  Toxicities were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0.
Time Frame: Baseline up to the end of Cycle 1 (each cycle=3 weeks)
Population: Per-Protocol Analysis Set: All participants who started treatment and who did not have first cycle major treatment deviations.
Measure: Number; unit: participants
Groups:
- Figitumumab 10 mg/kg + Sunitinib 25 mg CDD: Figitumumab 10 mg/kg IV on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle on a CDD schedule. Dose escalation proceeded to the next cohort if 0/3 or 1/6 participants experienced a DLT.
- Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD: Figitumumab 10 mg/kg IV on Day 1 of each 3-week cycle plus sunitinib 37.5 mg oral capsule on Day 1 of each 3-week cycle on a CDD schedule until disease progression or unacceptable toxicity.
- Figitumumab 20 mg/kg + Sunitinib 25 mg CDD: Figitumumab 20 mg/kg IV on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle on a CDD schedule until disease progression or unacceptable toxicity.
- Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1: Figitumumab 20 mg/kg on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle with 2 weeks of CDD followed by 1 week off, until disease progression or unacceptable toxicity.
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Number analyzed (Participants) | 20 | 7 | 12 | 6
participants | 0 | 1 | 3 | 1

2. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events, by National Cancer Institute (NCI) Common Terminology Criteria (CTC) for Adverse Events Grade Version 3.0
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs are events occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. If the same participant in a given treatment had more than one occurrence in the same preferred term event category, only the worst CTCAE grade was reported. Severity grades were 0 (no change from normal or reference range), 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening or disabling), and 5 (death).
Time Frame: Baseline, Day 1 of every cycle, Days 8 and 15 of Cycle 1, up to end of treatment (28 days post last dose)
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Number analyzed (Participants) | 20 | 7 | 12 | 6
percentage of participants
  Any AEs, Grade 1 | 0.0 | 0.0 | 16.7 | 0.0
  Any AEs, Grade 2 | 20.0 | 28.6 | 8.3 | 0.0
  Any AEs, Grade 3 | 40.0 | 42.9 | 50.0 | 16.7
  Any AEs, Grade 4 | 10.0 | 14.3 | 8.3 | 0.0
  Any AEs, Grade 5 | 30.0 | 14.3 | 16.7 | 83.3
  Any AEs, Total | 100.0 | 100.0 | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants With Hematologic Laboratory Test Abnormality
Description: Percentage of participants with hematologic laboratory abnormalities of CTC severity grades 1, 2, 3, or 4 (grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=life-threatening or disabling).
Time Frame: Baseline, Day 1 of every cycle, Days 8 and 15 of Cycle 1, up to end of treatment (28 days post last dose)
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Number analyzed (Participants) | 20 | 7 | 12 | 6
percentage of participants
  Hemoglobin | 70.0 | 85.7 | 75.0 | 83.3
  Lymphocytes (Absolute) | 85.0 | 85.7 | 91.7 | 33.3
  Neutrophils (Absolute) | 40.0 | 71.4 | 16.7 | 16.7
  Platelets | 80.0 | 100.0 | 58.3 | 50.0
  White Blood Cells | 65.0 | 71.4 | 41.7 | 33.3

4. Secondary Outcome: Percentage of Participants With Blood Chemistry Laboratory Test Abnormality
Description: Percentage of participants with blood chemistry laboratory abnormalities of CTC severity grades 1, 2, 3, or 4 (grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=life-threatening or disabling).
Time Frame: Baseline, Day 1 of every cycle, Days 8 and 15 of Cycle 1, up to end of treatment (28 days post last dose)
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study medication; n=number of participants evaluable for this outcome measure, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Number analyzed (Participants) | 20 | 7 | 12 | 6
percentage of participants
  Alanine Aminotransferase (n=19, 7, 12 ,6) | 57.9 | 57.1 | 33.3 | 0.0
  Alkaline Phosphatase (n=19, 7, 12, 6) | 52.6 | 57.1 | 58.3 | 66.7
  Aspartate Aminotransferase (n=19, 7, 12, 6) | 63.2 | 71.4 | 66.7 | 16.7
  Bicarbonate (n=19, 7, 12, 6) | 26.3 | 71.4 | 16.7 | 33.3
  Total Bilirubin (n=19, 7, 12, 6) | 21.1 | 71.4 | 25.0 | 0.0
  Creatinine (n=19, 7, 12, 6) | 26.3 | 57.1 | 41.7 | 50.0
  Hypercalcemia (n=19, 7, 12, 6) | 0.0 | 14.3 | 16.7 | 0.0
  Hyperglycemia (n=19, 7, 12, 6) | 78.9 | 100.0 | 75.0 | 83.3
  Hyperkalemia (n=19, 7, 12, 6) | 5.3 | 14.3 | 16.7 | 33.3
  Hypermagnesemia (n=17, 7, 12, 6) | 5.9 | 0.0 | 8.3 | 16.7
  Hypernatremia (n=19, 7, 12, 6) | 5.3 | 0.0 | 0.0 | 16.7
  Hypoalbuminemia (n=19, 7, 12, 6) | 42.1 | 42.9 | 33.3 | 83.3
  Hypocalcemia (n=19, 7, 12, 6) | 47.4 | 57.1 | 33.3 | 50.0
  Hypokalemia (n=19, 7, 12, 6) | 15.8 | 28.6 | 8.3 | 16.7
  Hypomagnesemia (n=17, 7, 12, 6) | 23.5 | 71.4 | 25.0 | 33.3
  Hyponatremia (n=19, 7, 12, 6) | 57.9 | 42.9 | 50.0 | 66.7
  Hypophosphatemia (n=17, 7, 11, 6) | 23.5 | 57.1 | 18.2 | 0.0

5. Secondary Outcome: Plasma Concentration at the End of Infusion (Cendinf) of Figitumumab
Time Frame: 0.5 hour predose and 1 hour post-infusion on Day 1 of Cycles 1 and 4
Population: Pharmacokinetic (PK) Analysis Set: Participants who received all scheduled doses of both drugs and completed all required PK assessments in the dose expansion cohort (figitumumab 10 mg/kg + sunitinib 25 mg CDD); n=number of participants in the indicated cycle.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram/liter (mg/L)
Groups:
- Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion): Figitumumab 10 mg/kg IV on Day 1 of each 3-week cycle plus sunitinib 25 mg oral capsule on Day 1 of each 3-week cycle on a CDD schedule, until disease progression or unacceptable toxicity.
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 11
milligram/liter (mg/L)
  Cycle 1 (n=11) | 203.1 (27)
  Cycle 4 (n=4) | 256.3 (28)

6. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Figitumumab
Description: AUClast is the area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: 0.5 hour predose and 1 hour post-infusion on Days 1, 2, 4, 8, 15, and 22 of Cycles 1 and 4
Population: PK Analysis Set: Participants who received all scheduled doses of both drugs and completed all required PK assessments in the dose expansion cohort (figitumumab 10 mg/kg + sunitinib 25 mg CDD); n=number of participants in the indicated cycle.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram*hour/milliliter (mg*hr/mL)
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 8
milligram*hour/milliliter (mg*hr/mL)
  Cycle 1 (n=8) | 27320 (20)
  Cycle 4 (n=4) | 37850 (4)

7. Secondary Outcome: Area Under the Curve From Time Zero to Day 22 [AUC504] of Figitumumab
Description: AUC504 is the area under the plasma concentration versus time curve from time zero (predose) to Day 22, where Day 22 is the nominal time (504 hours) of the predose sample for the next cycle.
Time Frame: 0.5 hour predose and 504 hours (Day 22) post-infusion of Cycles 1 and 4
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*hr/mL
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 8
mg*hr/mL
  Cycle 1 (n=8) | 33800 (18)
  Cycle 4 (n=4) | 46960 (6)

8. Secondary Outcome: Plasma Decay Half-Life (t1/2) of Figitumumab
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0.5 hour predose and 1 hour post-infusion on Days 1, 2, 4, 8, and 15 of Cycles 1 and 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 8
hours
  Cycle 1 (n=8) | 245.0 (55.0)
  Cycle 4 (n=4) | 268.0 (75.6)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sunitinib
Time Frame: 0.5 hour predose and 2, 4, 6, 8, 12, and 24 hours postdose on Day 15 of Cycle 1
Population: PK Analysis Set: Participants who received all scheduled doses of both drugs and completed all required PK assessments in the dose expansion cohort (figitumumab 10 mg/kg + sunitinib 25 mg CDD).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 11
nanogram/milliliter (ng/mL) | 39.19 (38)

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Sunitinib
Time Frame: 0.5 hour predose and 2, 4, 6, 8, 12, and 24 hours postdose on Day 15 of Cycle 1
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 11
hours | 4.07 [2.00 to 24.0]

11. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours Postdose (AUC24) of Sunitinib
Description: AUC24 is the area under the plasma concentration versus time curve from time zero (predose) to 24 hours postdose (0 to 24).
Time Frame: 0.5 hour predose and 2, 4, 6, 8, 12, and 24 hours postdose on Day 15 of Cycle 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 11
nanogram*hour/milliliter (ng*hr/mL) | 786.8 (42)

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Sunitinib
Time Frame: 0.5 hour predose on Day 1 of Cycle 2
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 11
ng/mL | 28.27 (47)

13. Secondary Outcome: Plasma Concentration at 24 Hours Postdose (C24) of Sunitinib
Time Frame: 24 hours postdose on Day 15 of Cycle 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (Dose Expansion)
Number analyzed (Participants) | 11
ng/mL | 28.87 (53)

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA)
Description: Assays for ADA assessment specific for figitumumab would have provided information regarding an immune response to the compound.
Time Frame: 0.5 hour pre-infusion on Day 1 in Cycles 1 and 2, at end of treatment, and during the last scheduled follow-up visit (5 months from the last dose of study drug)
Population: ADA Analysis Set: Participants who started treatment with study medication and provided at least 1 on-study ADA sample. Due to early termination of the study, ADA samples were not assayed.
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Objective Response (OR)
Description: Objective response (OR) was based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. CR was the complete disappearance of all target and non-target disease, no new lesions, or the normalization of markers (if markers were being followed). PR was greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions, no unequivocal progression of non-target disease, no new lesions, or no reappearance of lesions after a CR. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Baseline, Day 15 of every 2 cycles until disease progression up to follow-up (approximately 28 days following the last dose of study drug)
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Number analyzed (Participants) | 20 | 7 | 12 | 6
participants
  Complete Response (CR) | 0 | 0 | 0 | 0
  Partial Response (PR) | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1
Serious Adverse Events (participants affected / at risk) | 10/20 | 3/7 | 6/12 | 5/6
Other Adverse Events (participants affected / at risk) | 20/20 | 7/7 | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (N=20) | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD (N=7) | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD (N=12) | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1 (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Disease progression (General disorders) | 5 | 0 | 2 | 3
Pain (General disorders) | 2 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 10 mg/kg + Sunitinib 25 mg CDD (N=20) | Figitumumab 10 mg/kg + Sunitinib 37.5 mg CDD (N=7) | Figitumumab 20 mg/kg + Sunitinib 25 mg CDD (N=12) | Figitumumab 20 mg/kg + Sunitinib 25 mg Schedule 2/1 (N=6)
Anaemia (Blood and lymphatic system disorders) | 7 | 5 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 6 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 5 | 7 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 4 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 3 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 4 | 1
Asthenia (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 14 | 6 | 9 | 5
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 0
Mucosal dryness (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 4 | 3 | 2 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 2 | 0
Performance status decreased (General disorders) | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 3 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 0
Blood testosterone decreased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Pulmonary arterial pressure increased (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 3 | 3 | 0 | 0
Weight decreased (Investigations) | 2 | 2 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 12 | 4 | 3 | 0
Headache (Nervous system disorders) | 0 | 3 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 3 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Vaginal disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 7 | 3 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Debridement (Surgical and medical procedures) | 0 | 1 | 0 | 0
Skin graft (Surgical and medical procedures) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 2 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated prematurely. Subsequently, ADA samples were not assayed and the pharmacokinetics of sunitinib plus its metabolite were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.